CLINICAL TRIAL: NCT04874363
Title: The Effects of Smoking on Mortality in Intensive Care Unit in Patients With Acute Respiratory Syndrome Coronavirus 2 Infection
Brief Title: The Effects of Smoking on Mortality in Patients With Acute Respiratory Syndrome Coronavirus 2 Infection
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyhan Metin, medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 2810
Record Dates: First submitted 2021-05-01; First posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Covid19; Smoking
MeSH Terms: conditions — COVID-19; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- smoker: active smokers
  Interventions: Other: no intervention
- non-smoker: Patients who have never smoked
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This is a retrospective single centered study that was done in the ICU on patients with Covid-19 between 16th of March -16th of May in 2020 Retrospective records will be examined by examining the electronic data files of the patients.

There were two groups as smoker and non-smoker.

DETAILED DESCRIPTION:
The aims of the present study is to see the effects of smoking prevalence, the length of stay regarding the usage of cigarettes, and the effects on the mortality of COVID-19 in our intensive care unit(ICU).

This is a retrospective single centered study that was done in the ICU on patients with Covid-19 between 16th of March -16th of May in 2020. The demographic data, comorbidity status, the units they were accepted from, clinical symptoms , respiratory support, prevalence of smoking, length of stay in the ICU and mortalities of the patients weill be recorded. There are two groups as smoker and non-smoker.

ELIGIBILITY:
Inclusion Criteria:

* All the patient's data are diagnosed with acute respiratory syndrome Covid-19 over 18 years old

Exclusion Criteria:

* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Conditions regarded to the usage of cigarettes will be recorded as patients who are active smokers and patients who do not smoke.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Mortality | 3 months
  Mortality rates of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided